CLINICAL TRIAL: NCT01786707
Title: Phase 2 Study of Autologous Stem Cell and Hyperbaric Oxygen Therapy in Type 2 Diabetes Mellitus
Brief Title: Autologous Stem Cell and Hyperbaric Oxygen Therapy in Type 2 Diabetes Mellitus
Acronym: HOT
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Rodolfo Alejandro (Other)
Collaborators: Diabetes Research Institute Foundation (Other)
Responsible Party: Sponsor-Investigator, Rodolfo Alejandro, Director, Clinical Islet Transplant Program, Diabetes Research Institute, University of Miami
Organization: University of Miami (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 20070881
Record Dates: First submitted 2013-02-05; First posted 2013-02-08 (Estimated); Results first posted 2014-04-21 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2017-06

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: Type 2 Diabetes Mellitus; Hyperbaric oxygen therapy (HOT); Autologous Bone Marrow-Derived Buffy Coat; Stem cells (SC)
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Hyperbaric Oxygenation; Insulin; Metformin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Autologous SC and HOT (Experimental): Autologous stem cells and hyperbaric oxygen therapy
  Interventions: Biological: Autologous stem cells; Other: Hyperbaric oxygen therapy; Drug: Insulin; Drug: Metformin
- Control group (Active Comparator): Patients in a control group will continue with standard medical treatment (Insulin and Metformin)
  Interventions: Drug: Insulin; Drug: Metformin

INTERVENTIONS:
Biological: Autologous stem cells — Pancreatic artery infusion of Autologous Stem cells.
  Arms: Autologous SC and HOT
Other: Hyperbaric oxygen therapy
  Arms: Autologous SC and HOT
Drug: Insulin — Insulin dose as per clinical management
Drug: Metformin — Metformin dose as tolerated

SUMMARY:
A prospective, open labeled, randomized controlled clinical trial comparing the benefit of both hyperbaric oxygen therapy and intrapancreatic stem cell infusion to standard medical treatment alone for type 2 diabetes mellitus. Subjects will receive standard medical treatment (SMT) with insulin and metformin for 4 months (evaluation phase). Then they will be randomized into either the intervention group or the control group:

DETAILED DESCRIPTION:
This is a phase I/II, prospective, randomized case controlled study in patients with Type 2 Diabetes Mellitus (T2DM) that seeks to investigate whether the combination of intrapancreatic Autologous Stem Cell infusion (ASC) and Hyperbaric Oxygen treatment (HBO) can improve glycemic control and pancreatic function in T2DM patients compared to controls receiving standard medical treatment (SMT) with metformin and insulin alone.

New therapies that lead to stopping ß-cell damage and possible ß-cell regeneration may decrease the incidence and progression of T2DM chronic complications and together with achievable life style changes may improve general health and quality of life of T2DM patients. Preliminary data from a pilot study involving 25 subjects with T2DM that underwent a combined treatment using ASC+HBO showed a significant progressive and consistent reduction in plasma glucose and HbA1c with an increase in C-peptide in conjunction with a decrease in the number and dose of oral agents and/or insulin. These encouraging preliminary results require confirmation in a controlled, randomized prospective trial.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female patients age 45 to 65 years of age.
2. Ability to provide written informed consent.
3. Mentally stable and able to comply with the procedures of the study protocol.
4. Clinical history compatible with type 2 diabetes as defined by the Expert Committee on the Diagnosis and classification of Diabetes Mellitus.
5. Onset of Type 2 DM disease at 40 years of age.
6. T2DM duration: 2-15 years at the time of enrollment.
7. Basal C-peptide: 0.3 ng/mL
8. HbA1c of 7.5-12.5% before standard medical therapy. Patients must have been treated with SMT for minimum of 4 months prior to randomization. Insulin and metformin doses should be stable over the 3 months prior to randomization.
9. HbA1c: 7.5-9.5% at time of randomization.
10. Total insulin daily dose at baseline and at randomization <100 units/day.

Exclusion Criteria:

1. BMI >40 kg/m2.
2. Insulin requirements of >100 U/day, and HbA1c >9.5%
3. C-reactive protein >10.00
4. Uncontrolled blood pressure: Systolic Blood Pressure >140 mmHg or Diastolic Blood Pressure >80 mmHg Evidence of renal dysfunction, serum creatinine > 1.5 mg/dl (males) and 1.4 mg/dl (females)
5. Proteinuria >300 mg/day
6. History or EKG evidence of myocardial infarction or any degree of heart failure
7. Female participants: Positive pregnancy test, presently breast-feeding, or unwillingness to use effective contraceptive measures for the duration of the study. Male participants: intent to procreate 3 months before or after the intervention or unwillingness to use effective measures of contraception.
8. Active infection including hepatitis B, hepatitis C, HIV, or Tuberculosis. Positive tests are acceptable only if associated with a history of previous vaccination in the absence of any sign of active infection.
9. Known active alcohol or substance abuse including cigarette/cigar smoking
10. Baseline Hgb below the lower limits of normal at the local laboratory; lymphopenia (<1,000/L), neutropenia (<1,500/L), or thrombocytopenia (platelets <100,000/L).
11. A history of Factor V deficiency or other coagulopathy defined by International normalized ratio (INR) >1.5, Partial thromboplastin time (PTT) >40, Prothrombin time (PT) >15.
12. Acute or chronic pancreatitis.
13. Symptomatic peptic ulcer disease.
14. Hyperlipidemia despite medical therapy
15. Receiving treatment for a medical condition requiring chronic use of systemic corticosteroids in the past six months.
16. Symptomatic cholecystolithiasis.
17. Use of any investigational agents within 4 weeks of enrollment.
18. Admission to hospital for any reason in the 14 days prior to enrollment.
19. History or presence of active proliferative diabetic retinopathy or macular edema.
20. Any malignancy.
21. Hepatic enzyme levels upper normal limits.
22. Total bilirubin upper normal limits unless secondary to known benign condition.
23. Abdominal aortic aneurysm.
24. History of cerebro-vascular accident.
25. Any patient with acute or subacute decompensation from diabetes.
26. Any acute or chronic infectious condition that in the criteria of the investigator would be a risk for the patient.
27. Hypoproteinemia, cachexia or terminal states; history of anorexia/bulimia; respiratory insufficiency; history of chronic sinusitis (sinusitis lasting more than 8 weeks in the past year) or recurrent acute sinusitis (sinusitis lasting more than 4 weeks more than four times in the past year.
28. Any contraindication to hyperbaric oxygen treatment.
29. Subjects treated with any medication that could interfere with the outcome of the study.
30. Subjects positive for auto-antibodies
31. History of Cushing syndrome (endogenous or iatrogenic).
32. History of allergy to iodine or iodinated materials.
33. Abnormal thyroid function
34. Any medical condition that, in the opinion of the investigator, will interfere with the safe completion of the trial.

Ages: 45 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2009-07; Primary Completion 2011-03 (Actual); Study Completion 2013-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rodolfo Alejandro, MD, Principal Investigator — Diabetes Research Institute, University of Miami Miller School of Medicine
Locations (1):
- Diabetes Research Institute, University of Miami Miller School of Medicine, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Autologous Stem Cell and HOT: Autologous stem cells (SC) and hyperbaric oxygen therapy
  Autologous stem cells and hyperbaric oxygen therapy: Subjects will receive standard medical treatment (SMT) with insulin and metformin for 4 months. Then they will be randomized to either control or intervention groups. HOT and SC group: combination of HOT therapy and intrapancreatic autologous SC infusion in addition to SMT.
- Control Group: Patients in a control group will continue with standard medical treatment (SMT)
Period: Overall Study
Arm/Group | Autologous Stem Cell and HOT | Control Group
Started | 1 | 1
Completed | 0 | 0
Not Completed | 1 | 1
Not completed — Lost to Follow-up | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Autologous SC and HOT: Autologous stem cells and hyperbaric oxygen therapy
  Autologous stem cells and hyperbaric oxygen therapy: Subjects will receive standard medical treatment (SMT) with insulin and metformin for 4 months. Then they will be randomized to either control or intervention groups. HOT and SC group: combination of HOT therapy and intrapancreatic autologous SC infusion in addition to SMT.
- Total: Total of all reporting groups
Arm/Group | Autologous SC and HOT | Control Group | Total
Number analyzed (Participants) | 1 | 1 | 2
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 1 | 1 | 2
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 1 | 1
  Male | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With a Reduction of HbA1c of >0.5%
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Autologous SC and HOT | Control Group
Number analyzed (Participants) | 1 | 1
Participants | 0 | 0

2. Secondary Outcome: The Number of Subjects With a Reduction of >1% in HbA1c
Time Frame: at 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Autologous SC and HOT | Control Group
Number analyzed (Participants) | 1 | 1
Participants | 0 | 0

ADVERSE EVENTS:
Arm/Group | Autologous SC and HOT | Control Group
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/1
Other Adverse Events (participants affected / at risk) | 0/1 | 0/1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes